CLINICAL TRIAL: NCT03541369
Title: A Phase 1 First-In-Human Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Efficacy of AMG 427 in Subjects With Relapsed/Refractory Acute Myeloid Leukemia.
Brief Title: Safety, Tolerability, PK, PD, and Efficacy of AMG 427 in Subjects With Relapsed/Refractory Acute Myeloid Leukemia
Acronym: 20170528
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Premature discontinuation of study, a strategic decision.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20170528; BB-IND 138440 (Other Grant/Funding Number: IND Number); 2018-001389-40 (EudraCT Number)
Record Dates: First submitted 2018-05-18; First posted 2018-05-30 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-07

CONDITIONS: Relapsed/Refractory Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation Phase (Experimental): AMG 427 Dose-finding phase of the study
  Interventions: Drug: AMG 427
- Dose Expansion Phase (Experimental): AMG 427 MTD identified in dose escalation phase (or lower) will be administered to subjects.
  Interventions: Drug: AMG 427

INTERVENTIONS:
Drug: AMG 427 — AMG 427 will be administered as an intravenous (IV) infusion in adult subjects with relapsed/refractory AML.
  Other Names: AMG 427; 20170528

SUMMARY:
Evaluate the safety and tolerability of AMG 427 in adult subjects with relapsed/refractory (R/R) acute myeloid leukemia (AML). Estimate the maximum tolerated dose (MTD) and / or a biologically optimal dose (eg, recommended phase 2 dose [RP2D]).

DETAILED DESCRIPTION:
Evaluate the safety and tolerability of AMG 427 in adult subjects with relapsed/refractory AML. Estimate the maximum tolerated dose (MTD) and / or a biologically optimal dose (eg, recommended phase 2 dose [RP2D]). Approximately 80 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent prior to initiation of any study-specific activities/procedures.
* Subjects greater than or equal to 18 years of age at the time of signing consent.
* For relapsed/refractory AML subjects only, AML as defined by the WHO Classification as persisting or recurring following 1 or more treatment courses (exceptions noted in exclusion criteria).
* Myeloblasts greater than or equal to 5% in bone marrow, as confirmed by immunophenotype by flow cytometry.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of less than or equal to 2.
* Renal function as follows: serum creatinine less than 2.0 mg/dL (176.84 µmol/L); estimated glomerular filtration rate (eGFR) greater than 30 mL/min/1.73 m^2.
* Hepatic function as follows: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 3.0 x upper limit of normal (ULN); bilirubin less than or equal to 1.5 x ULN (unless considered due to Gilbert's syndrome or hemolysis).
* No active tuberculosis in the setting of anti-tumor necrosis factor (TNF) therapy - National guidelines should be followed for the appropriate tuberculosis screening in the setting of anti-TNF therapy, including a minimum of:

  * Subject has a negative test for tuberculosis during screening defined as either:

    * Negative purified protein derivative (PPD) (< 5 mm induration at 48 to 72 hours after test is placed) OR
    * Negative Quantiferon test
  * Subjects with positive PPD and a history of bacillus Calmette-Guérin vaccination are allowed with a negative Quantiferon test.
  * Subjects with a positive PPD test (without a history of bacillus Calmette-Guérin vaccination) or subjects with a positive or indeterminate Quantiferon test are allowed if they have all of the following:

    * No symptoms, per tuberculosis worksheet provided by Amgen
    * Documented history of a completed course of adequate treatment or prophylaxis (per local standard of care) prior to the start of investigational product
    * No known exposure to a case of active tuberculosis after most recent prophylaxis
    * No evidence of active tuberculosis on chest radiograph within 3 months prior to the first dose of investigational product (substudy subjects only)

Exclusion Criteria:

* Patients with acute promyelocytic leukemia (APML).
* Active extramedullary AML in the central nervous system (CNS)
* Known hypersensitivity to immunoglobulins.
* White blood cells (WBC) greater than 15,000 cells/mcL (15 cells x 10^9/L) at screening (hydroxyurea is permitted to enable eligibility).
* Subjects with a prior or concurrent malignancy whose natural history or treatment is anticipated to interfere with the safety or efficacy assessment of the investigational regimen. Exception: Subjects with prior or concurrent malignancy not anticipated to interfere with the safety or efficacy of the investigational regimen may be included only after discussion with the Amgen Medical Monitor.
* Autologous hematopoietic stem cell transplant (HSCT) within 6 weeks prior to start of AMG 427 treatment.
* Allogeneic HSCT within 3 months prior to start of AMG 427 treatment.
* Any graft-versus-host disease requiring systemic therapy with immunomodulators.
* History or evidence of significant cardiovascular risk including any of the following: symptomatic congestive heart failure, unstable angina, clinically significant arrhythmias (eg, ventricular fibrillation, ventricular tachycardia etc.), recent coronary angioplasty, intra-cardiac defibrillators or any clinically relevant concurrent disorder that may pose a risk to subject safety or interfere with study evaluation, procedures, or completion.
* History of arterial thrombosis (eg, stroke or transient ischemic attack) in the past 3 months.
* Active infection requiring intravenous antibiotics within 1 week of study enrollment (day 1). Antibiotics may be administered for prophylaxis as per institutional standards up to and after enrollment.
* Known positive test for human immunodeficiency virus (HIV).
* Positive for hepatitis B surface antigen (HepBsAg).
* Positive for hepatitis C or chronic hepatitis C. Possible exceptions: acute hepatitis C and completely cleared of the virus (demonstrated by negative viral load), chronic hepatitis C with undetectable viral load defined by sustained virologic response 24 weeks (SVR24) after completion of anti-hepatitis C treatment.
* Live vaccination(s) within 4 weeks before the start of AMG 427 treatment on day 1, during treatment, and until the end of the last study dose.
* Unresolved toxicities from prior antitumor therapy, defined as not having resolved to Common Terminology Criteria for Adverse Events (CTCAE), version 4.0 grade 1 (with the exception of myelosuppression, eg, neutropenia, anemia, thrombocytopenia), or to levels dictated in the eligibility criteria with the exception of alopecia or toxicities from prior antitumor therapy that are considered irreversible (defined as having been present and stable for greater than 2 months) which may be allowed if they are not otherwise described in the exclusion criteria AND there is agreement to allow by both the investigator and sponsor.
* Antitumor therapy (chemotherapy, antibody therapy, molecular-targeted therapy, or investigational agent) within 14 days of day 1. Exception: hydroxyurea to control peripheral blood leukemic cell counts is allowed until start of investigational product treatment. Exception: antitumor therapies with short half-lives only require passing of 5 half-lives from last dose, and after discussion with sponsor.
* Treatment with systemic immune modulators including, but not limited to, non-topical systemic corticosteroids, cyclosporine, and tacrolimus within 2 weeks before enrollment (day 1). Exceptions: physiologic replacement steroids or steroids for treatment of transfusion/hypersensitivity reactions.
* Prior treatment with a fms-like tyrosine kinase 3 (FLT3) targeting chimeric antigen receptor T cell (CAR-T)
* Major surgery within 28 days of study day 1 with the exception of biopsy and insertion of central venous catheter.
* History or evidence of any other clinically significant disorder, condition or disease that, in the opinion of the investigator or Amgen medical monitor would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.
* Males and females of reproductive potential who are unwilling to practice a highly effective method(s) of birth control while on study through 4 weeks after receiving the last dose of study drug. Acceptable methods of highly effective birth control include sexual abstinence (males, females); vasectomy; bilateral tubal ligation/occlusion; or a condom with spermicide (men) in combination with hormonal birth control or intrauterine device (IUD) (women).
* Females who are lactating/breastfeeding or who plan to breastfeed while on study through 4 weeks after receiving the last dose of study drug.
* Females with a positive pregnancy test.
* Females planning to become pregnant while on study through 4 weeks after receiving the last dose of study drug.
* Subjects likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures to the best of the subject's and investigator's knowledge.
* History of multiple sclerosis or any other demyelinating disease.
* No active hepatitis secondary to alcoholic hepatitis or nonalcoholic steatohepatitis.
* History or evidence of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection unless agreed upon with Medical Monitor and meeting the following criteria:

  * Negative test for SARS-CoV-2 RNA by reverse transcriptase-polymerase chain reaction (RT-PCR) within 72 hours of first dose of investigational product
  * No acute symptoms of coronavirus disease 2019 (COVID-19) disease within 10 days prior to first dose of investigational product (counted from day of positive test for asymptomatic subjects)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (16):
- United States (7):
  - City of Hope National Medical Center, Duarte, California
  - Northwestern University, Evanston, Illinois
  - Johns Hopkins, Baltimore, Maryland
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (2):
  - The Alfred Hospital, Melbourne, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
- University Health Network-Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- Germany (2):
  - Universitätsklinikum Carl Gustav Carus der Technischen Universität Dresden, Dresden
  - Klinikum der Universitaet Muenchen Campus Grosshadern, München
- Japan (2):
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - University of Fukui Hospital, Yoshida-gun, Fukui
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 11 study centers in 5 countries, including Australia, Canada, Germany, Japan, and the United States, and participated from 14 September 2018 to 21 February 2023.
Pre-assignment Details: Participants were enrolled into first-in-human (FIH) groups with no step dosing (cohorts 1 - 7a), and with step dosing (cohorts 7b - 13), into extended intravenous (eIV) groups (cohorts 14 -15), and into an etanercept substudy (cohorts 16 - 17). Dosing was from Dose A (lowest) to Dose M (highest).
Groups:
- Cohort 1 (FIH): Emirodatamab Dose A: Emirodatamab Dose A was administered as an intravenous (IV) infusion in a 2-week cycle with no step dosing. Dexamethasone 8 mg IV was administered within 1 hour before dosing.
- Cohort 2 (FIH): Emirodatamab Dose B: Emirodatamab Dose B was administered as an IV infusion in a 2-week cycle with no step dosing. Dexamethasone 8 mg IV was administered within 1 hour before dosing.
- Cohort 3 (FIH): Emirodatamab Dose C: Emirodatamab Dose C was administered as an IV infusion in a 2-week cycle with no step dosing. Dexamethasone 8 mg IV was administered within 1 hour before dosing.
- Cohort 4 (FIH): Emirodatamab Dose D: Emirodatamab Dose D was administered as an IV infusion in a 2-week cycle with no step dosing. Dexamethasone 8 mg IV was administered within 1 hour before dosing.
- Cohort 5 (FIH): Emirodatamab Dose E: Emirodatamab Dose E was administered as an IV infusion in a 2-week cycle with no step dosing. Dexamethasone 8 mg IV was administered within 1 hour before dosing.
- Cohort 6 (FIH): Emirodatamab Dose F: Emirodatamab Dose F was administered as an IV infusion in a 2-week cycle with no step dosing. Dexamethasone 8 mg IV was administered within 1 hour before dosing.
- Cohort 7a (FIH): Emirodatamab Dose G: Emirodatamab Dose G was administered as an IV infusion in a 2-week cycle with no step dosing. Dexamethasone 8 mg IV was administered within 1 hour before dosing.
- Cohort 7b (FIH): Emirodatamab Dose F/Dose G: Emirodatamab was administered as an IV infusion with step dosing; Dose F followed by Dose G (2-week cycle). Dexamethasone 8 mg IV was administered within 1 hour before dosing.
- Cohort 8 (FIH): Emirodatamab Dose F/Dose H: Emirodatamab was administered as an IV infusion with step dosing; Dose F followed by Dose H (2-week cycle). Dexamethasone 8 mg IV was administered within 1 hour before dosing.
- Cohort 9 (FIH): Emirodatamab Dose F/Dose H/Dose I: Emirodatamab was administered as an IV infusion with step dosing; Dose F followed by Doses H and I (2-week cycle). Dexamethasone 8 mg IV was administered within 1 hour before dosing.
- Cohort 10 (FIH): Emirodatamab Dose F/Dose H/Dose J: Emirodatamab was administered as an IV infusion with step dosing; Dose F followed by Doses H and J (2-week cycle). Dexamethasone 8 mg IV was administered within 1 hour before dosing.
- Cohort 11 (FIH): Emirodatamab Dose F/Dose H/Dose K: Emirodatamab was administered as an IV infusion with step dosing; Dose F followed by Doses H and K (2-week cycle). Dexamethasone 8 mg IV was administered within 1 hour before dosing.
- Cohort 12 (FIH): Emirodatamab Dose F/Dose H/Dose L: Emirodatamab was administered as an IV infusion with step dosing; Dose F followed by Doses H and L (2-week cycle). Dexamethasone 8 mg IV was administered within 1 hour before dosing.
- Cohort 13 (FIH): Emirodatamab Dose F/Dose H/Dose M: Emirodatamab was administered as an IV infusion with step dosing; Dose F followed by Doses H and M (2-week cycle). Dexamethasone 8 mg IV was administered within 1 hour before dosing.
- Cohort 14 (eIV): Emirodatamab Dose F/Dose H/Dose J/Dose K: Emirodatamab was administered as an eIV infusion with step dosing; Dose F followed by Doses H, J, and K (2-week cycle). Dexamethasone 8 mg IV was administered within 1 hour before dosing.
- Cohort 15 (eIV): Emirodatamab Dose F/Dose H/Dose J: Emirodatamab was administered as an eIV infusion with step dosing; Dose F followed by Doses H and J (2-week cycle). Dexamethasone 8 mg IV was administered within 1 hour before dosing.
- Cohort 16: Etanercept + Emirodatamab Dose E: Emirodatamab Dose E was administered as an IV infusion in a 2-week cycle. Participants were administered etanercept 50 mg subcutaneously (SC) 2 days before emirodatamab dosing. Dexamethasone 8 mg IV was administered within 1 hour before emirodatamab dosing.
- Cohort 17: Etanercept + Emirodatamab Dose F: Emirodatamab Dose F was administered as an IV infusion in a 2-week cycle. Participants were administered etanercept 50 mg SC 2 days before emirodatamab dosing. Dexamethasone 8 mg IV was administered within 1 hour before emirodatamab dosing.
Period: Overall Study
Arm/Group | Cohort 1 (FIH): Emirodatamab Dose A | Cohort 2 (FIH): Emirodatamab Dose B | Cohort 3 (FIH): Emirodatamab Dose C | Cohort 4 (FIH): Emirodatamab Dose D | Cohort 5 (FIH): Emirodatamab Dose E | Cohort 6 (FIH): Emirodatamab Dose F | Cohort 7a (FIH): Emirodatamab Dose G | Cohort 7b (FIH): Emirodatamab Dose F/Dose G | Cohort 8 (FIH): Emirodatamab Dose F/Dose H | Cohort 9 (FIH): Emirodatamab Dose F/Dose H/Dose I | Cohort 10 (FIH): Emirodatamab Dose F/Dose H/Dose J | Cohort 11 (FIH): Emirodatamab Dose F/Dose H/Dose K | Cohort 12 (FIH): Emirodatamab Dose F/Dose H/Dose L | Cohort 13 (FIH): Emirodatamab Dose F/Dose H/Dose M | Cohort 14 (eIV): Emirodatamab Dose F/Dose H/Dose J/Dose K | Cohort 15 (eIV): Emirodatamab Dose F/Dose H/Dose J | Cohort 16: Etanercept + Emirodatamab Dose E | Cohort 17: Etanercept + Emirodatamab Dose F
Started | 1 | 1 | 1 | 1 | 5 | 4 | 2 | 3 | 4 | 4 | 4 | 4 | 7 | 3 | 7 | 3 | 6 | 4
Completed | 1 | 1 | 1 | 0 | 3 | 1 | 1 | 0 | 0 | 2 | 3 | 3 | 2 | 0 | 3 | 1 | 1 | 0
Not Completed | 0 | 0 | 0 | 1 | 2 | 3 | 1 | 3 | 4 | 2 | 1 | 1 | 5 | 3 | 4 | 2 | 5 | 4
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 2 | 1 | 0 | 2 | 1 | 1 | 1 | 0 | 1
Not completed — Decision by sponsor | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 4 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1 (FIH): Emirodatamab Dose A: Emirodatamab Dose A was administered as an IV infusion in a 2-week cycle with no step dosing. Dexamethasone 8 mg IV was administered within 1 hour before dosing.
- Cohort 16: Etanercept + Emirodatamab Dose E: Emirodatamab Dose E was administered as an IV infusion in a 2-week cycle. Participants were administered etanercept 50 mg SC 2 days before emirodatamab dosing. Dexamethasone 8 mg IV was administered within 1 hour before emirodatamab dosing.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (FIH): Emirodatamab Dose A | Cohort 2 (FIH): Emirodatamab Dose B | Cohort 3 (FIH): Emirodatamab Dose C | Cohort 4 (FIH): Emirodatamab Dose D | Cohort 5 (FIH): Emirodatamab Dose E | Cohort 6 (FIH): Emirodatamab Dose F | Cohort 7a (FIH): Emirodatamab Dose G | Cohort 7b (FIH): Emirodatamab Dose F/Dose G | Cohort 8 (FIH): Emirodatamab Dose F/Dose H | Cohort 9 (FIH): Emirodatamab Dose F/Dose H/Dose I | Cohort 10 (FIH): Emirodatamab Dose F/Dose H/Dose J | Cohort 11 (FIH): Emirodatamab Dose F/Dose H/Dose K | Cohort 12 (FIH): Emirodatamab Dose F/Dose H/Dose L | Cohort 13 (FIH): Emirodatamab Dose F/Dose H/Dose M | Cohort 14 (eIV): Emirodatamab Dose F/Dose H/Dose J/Dose K | Cohort 15 (eIV): Emirodatamab Dose F/Dose H/Dose J | Cohort 16: Etanercept + Emirodatamab Dose E | Cohort 17: Etanercept + Emirodatamab Dose F | Total
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 5 | 4 | 2 | 3 | 4 | 4 | 4 | 4 | 7 | 3 | 7 | 3 | 6 | 4 | 64
Age, Customized [Count of Participants; unit: Participants]
  18 - 64 years | 1 | 1 | 1 | 1 | 3 | 3 | 2 | 2 | 3 | 3 | 4 | 3 | 5 | 2 | 3 | 2 | 3 | 1 | 43
  65 - 74 years | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 1 | 4 | 1 | 2 | 3 | 18
  75 - 84 years | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
  ≥ 85 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 1 | 2 | 2 | 5 | 3 | 3 | 0 | 2 | 2 | 27
  Male | 0 | 0 | 1 | 1 | 3 | 3 | 2 | 2 | 3 | 3 | 2 | 2 | 2 | 0 | 4 | 3 | 4 | 2 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 7
  Not Hispanic or Latino | 1 | 1 | 1 | 1 | 4 | 3 | 2 | 3 | 3 | 3 | 4 | 4 | 6 | 3 | 5 | 2 | 6 | 4 | 56
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 1 | 1 | 0 | 12
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 1 | 0 | 0 | 1 | 2 | 2 | 1 | 2 | 4 | 3 | 3 | 2 | 5 | 3 | 6 | 2 | 5 | 3 | 45
  Other | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Dose Limiting Toxicity (DLT)
Description: A DLT was any of the following during the DLT window, assessed by Common Terminology Criteria for Adverse Events (CTCAE) v 4.0 except for cytokine release syndrome (CRS) grading:
  * drug-induced liver injury
  * any treatment-related death
  * Grade 2 CRS not resolving to ≤ grade 1 within 7 days; grade 3 CRS not resolving to ≤ grade 1 within 7 days; grade 3 CRS reported at the initial run-in dose; 2 separate grade 3 CRS events
  * Grade 4 CRS/infusion reactions
  * Grade 3-5 non-hematologic toxicity not clearly resulting from underlying leukemia except: alopecia, grade 3 rash, fatigue, asthenia, fever, anorexia, or constipation, nausea, vomiting or diarrhea not requiring tube feeding, total parenteral nutrition, or requiring/prolonging hospitalization; infection, bleeding, or other expected complication of cytopenias due to underlying leukemia; grade 3 infusion reaction including CRS; grade 3 tumor lysis syndrome
  * Grade 4 neutropenia persisting beyond 42 days in absence of leukemia.
Time Frame: Days 1 to 28 for each cohort (28 days)
Population: The DLT evaluable set included all DLT-evaluable participants, defined as participants who received the doses planned for the respective cohort, and completed the DLT window of 28 days for all cohorts unless they dropped out before completion of the DLT window for reasons other than a DLT. Exception: participant had received the planned doses in cycle 1 and dropped out within 1 week of the completion of the DLT period due to progressive disease, that participant was considered DLT-evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (FIH): Emirodatamab Dose A | Cohort 2 (FIH): Emirodatamab Dose B | Cohort 3 (FIH): Emirodatamab Dose C | Cohort 4 (FIH): Emirodatamab Dose D | Cohort 5 (FIH): Emirodatamab Dose E | Cohort 6 (FIH): Emirodatamab Dose F | Cohort 7a (FIH): Emirodatamab Dose G | Cohort 7b (FIH): Emirodatamab Dose F/Dose G | Cohort 8 (FIH): Emirodatamab Dose F/Dose H | Cohort 9 (FIH): Emirodatamab Dose F/Dose H/Dose I | Cohort 10 (FIH): Emirodatamab Dose F/Dose H/Dose J | Cohort 11 (FIH): Emirodatamab Dose F/Dose H/Dose K | Cohort 12 (FIH): Emirodatamab Dose F/Dose H/Dose L | Cohort 13 (FIH): Emirodatamab Dose F/Dose H/Dose M | Cohort 14 (eIV): Emirodatamab Dose F/Dose H/Dose J/Dose K | Cohort 15 (eIV): Emirodatamab Dose F/Dose H/Dose J | Cohort 16: Etanercept + Emirodatamab Dose E | Cohort 17: Etanercept + Emirodatamab Dose F
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 4 | 3 | 2 | 3 | 3 | 3 | 3 | 4 | 7 | 2 | 7 | 3 | 5 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2

2. Primary Outcome: Number of Participants Who Experienced Treatment-emergent Adverse Events (TEAEs) and Treatment-related TEAEs
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical trial participant.
  A TEAE was an AE that started on or after the first dose of investigational product (emirodatamab) up to 30 days after the end of investigational product or end of study date, whichever was earlier.
  A treatment-related AE was any TEAE that per investigator review had a reasonable possibility of being caused by the investigational product (emirodatamab).
Time Frame: Day 1 Cycle 1 to 30 days after last dose of investigational product or end of study; median treatment duration was 0.62 months
Population: For Cohorts 1-15, the safety analysis set included all participants who received at least 1 dose of emirodatamab. For cohorts 16 and 17, the safety analysis set included all participants who received at least 1 dose of emirodatamab or etanercept.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (FIH): Emirodatamab Dose A | Cohort 2 (FIH): Emirodatamab Dose B | Cohort 3 (FIH): Emirodatamab Dose C | Cohort 4 (FIH): Emirodatamab Dose D | Cohort 5 (FIH): Emirodatamab Dose E | Cohort 6 (FIH): Emirodatamab Dose F | Cohort 7a (FIH): Emirodatamab Dose G | Cohort 7b (FIH): Emirodatamab Dose F/Dose G | Cohort 8 (FIH): Emirodatamab Dose F/Dose H | Cohort 9 (FIH): Emirodatamab Dose F/Dose H/Dose I | Cohort 10 (FIH): Emirodatamab Dose F/Dose H/Dose J | Cohort 11 (FIH): Emirodatamab Dose F/Dose H/Dose K | Cohort 12 (FIH): Emirodatamab Dose F/Dose H/Dose L | Cohort 13 (FIH): Emirodatamab Dose F/Dose H/Dose M | Cohort 14 (eIV): Emirodatamab Dose F/Dose H/Dose J/Dose K | Cohort 15 (eIV): Emirodatamab Dose F/Dose H/Dose J | Cohort 16: Etanercept + Emirodatamab Dose E | Cohort 17: Etanercept + Emirodatamab Dose F
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 5 | 4 | 2 | 3 | 4 | 4 | 4 | 4 | 7 | 3 | 7 | 3 | 6 | 4
Participants
  TEAEs | 1 | 1 | 1 | 1 | 5 | 4 | 2 | 3 | 4 | 4 | 4 | 4 | 7 | 3 | 7 | 3 | 6 | 4
  Treatment-related TEAEs | 1 | 1 | 1 | 1 | 5 | 4 | 2 | 3 | 4 | 4 | 4 | 4 | 6 | 3 | 7 | 3 | 6 | 2

3. Secondary Outcome: Maximum Observed Concentration (Cmax) of Emirodatamab
Description: Serum concentrations of emirodatamab were determined using a validated assay. Noncompartmental analysis was performed for estimation of pharmacokinetic (PK) parameters. Concentrations below the LLOQ (0.05 ng/mL) were set to zero before data analysis.
Time Frame: Cohorts 1, 2, 3, 4, 5, 6, 7a, 7b, 8, 9, 10, 11, 12, 13, 16 and 17: Cycle 1 Day 5 (C1D5); Cohorts 14 and 15: Cycle 1 Day 8 (C1D8) (sampling pre-dose up to 72 hours post-dose)
Population: The PK analysis set included all participants who received at least 1 dose of the investigational product and had at least 1 PK sample collected. Participants were included for PK analysis unless the number of data points required for analysis was not enough, or significant protocol deviations had affected the data, or if key dosing or sampling information is missing. Participants with data available at each timepoint are presented.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Cohort 1 (FIH): Emirodatamab Dose A | Cohort 2 (FIH): Emirodatamab Dose B | Cohort 3 (FIH): Emirodatamab Dose C | Cohort 4 (FIH): Emirodatamab Dose D | Cohort 5 (FIH): Emirodatamab Dose E | Cohort 6 (FIH): Emirodatamab Dose F | Cohort 7a (FIH): Emirodatamab Dose G | Cohort 7b (FIH): Emirodatamab Dose F/Dose G | Cohort 8 (FIH): Emirodatamab Dose F/Dose H | Cohort 9 (FIH): Emirodatamab Dose F/Dose H/Dose I | Cohort 10 (FIH): Emirodatamab Dose F/Dose H/Dose J | Cohort 11 (FIH): Emirodatamab Dose F/Dose H/Dose K | Cohort 12 (FIH): Emirodatamab Dose F/Dose H/Dose L | Cohort 13 (FIH): Emirodatamab Dose F/Dose H/Dose M | Cohort 14 (eIV): Emirodatamab Dose F/Dose H/Dose J/Dose K | Cohort 15 (eIV): Emirodatamab Dose F/Dose H/Dose J | Cohort 16: Etanercept + Emirodatamab Dose E | Cohort 17: Etanercept + Emirodatamab Dose F
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 4 | 3 | 1 | 3 | 3 | 4 | 3 | 3 | 5 | 3 | 6 | 2 | 5 | 1
ng/mL
  C1D5 Free Emirodatamab: number analyzed (Participants) | 1 | 1 | 1 | 1 | 4 | 3 | 1 | 3 | 3 | 4 | 3 | 3 | 5 | 3 | 0 | 0 | 5 | 1
  C1D5 Free Emirodatamab | 0.0963 [0.0963 to 0.0963] | 0.00 [0.00 to 0.00] | 0.116 [0.116 to 0.116] | 0.0879 [0.0879 to 0.0879] | 1.38 [0.909 to 5.19] | 1.10 [0.665 to 7.15] | 2.72 [2.72 to 2.72] | 7.54 [2.63 to 42.3] | 14.1 [3.57 to 28.4] | 21.4 [8.47 to 77.2] | 124 [11.5 to 137] | 29.7 [17.3 to 180] | 156 [13.7 to 355] | 46.7 [23.3 to 276] |  |  | 0.487 [0.115 to 2.38] | 0.838 [0.838 to 0.838]
  C1D8 Free Emirodatamab: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2 | 0 | 0
  C1D8 Free Emirodatamab |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 161 [4.92 to 232] | 36.7 [13.0 to 60.4] |  |

4. Secondary Outcome: Time to Reach Cmax (Tmax) of Emirodatamab
Description: Serum concentrations of emirodatamab were determined using a validated assay. Noncompartmental analysis was performed for estimation of PK parameters. Concentrations below the LLOQ (0.05 ng/mL) were set to zero before data analysis.
Time Frame: Cohorts 1, 2, 3, 4, 5, 6, 7a, 7b, 8, 9, 10, 11, 12, 13, 16 and 17: C1D5; Cohorts 14 and 15: C1D8 (sampling pre-dose up to 72 hours post-dose)
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1 (FIH): Emirodatamab Dose A | Cohort 2 (FIH): Emirodatamab Dose B | Cohort 3 (FIH): Emirodatamab Dose C | Cohort 4 (FIH): Emirodatamab Dose D | Cohort 5 (FIH): Emirodatamab Dose E | Cohort 6 (FIH): Emirodatamab Dose F | Cohort 7a (FIH): Emirodatamab Dose G | Cohort 7b (FIH): Emirodatamab Dose F/Dose G | Cohort 8 (FIH): Emirodatamab Dose F/Dose H | Cohort 9 (FIH): Emirodatamab Dose F/Dose H/Dose I | Cohort 10 (FIH): Emirodatamab Dose F/Dose H/Dose J | Cohort 11 (FIH): Emirodatamab Dose F/Dose H/Dose K | Cohort 12 (FIH): Emirodatamab Dose F/Dose H/Dose L | Cohort 13 (FIH): Emirodatamab Dose F/Dose H/Dose M | Cohort 14 (eIV): Emirodatamab Dose F/Dose H/Dose J/Dose K | Cohort 15 (eIV): Emirodatamab Dose F/Dose H/Dose J | Cohort 16: Etanercept + Emirodatamab Dose E | Cohort 17: Etanercept + Emirodatamab Dose F
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 4 | 3 | 1 | 3 | 3 | 4 | 3 | 3 | 5 | 3 | 6 | 2 | 5 | 1
hours
  C1D5 Free Emirodatamab: number analyzed (Participants) | 1 | 1 | 1 | 1 | 4 | 3 | 1 | 3 | 3 | 4 | 3 | 3 | 5 | 3 | 0 | 0 | 5 | 1
  C1D5 Free Emirodatamab | 1.2 [1.2 to 1.2] | 0.00 [0.00 to 0.00] | 5.9 [5.9 to 5.9] | 2.0 [2.0 to 2.0] | 1.0 [0.88 to 2.2] | 1.1 [1.1 to 2.0] | 1.9 [1.9 to 1.9] | 1.1 [1.0 to 1.1] | 1.6 [1.0 to 1.6] | 2.5 [1.6 to 2.6] | 1.7 [1.5 to 2.5] | 1.8 [1.6 to 2.6] | 1.9 [1.6 to 2.6] | 2.4 [1.6 to 2.7] |  |  | 1.3 [1.1 to 2.6] | 1.8 [1.8 to 1.8]
  C1D8 Free Emirodatamab: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2 | 0 | 0
  C1D8 Free Emirodatamab |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 1.7 [1.5 to 1.8] | 1.9 [1.7 to 2.1] |  |

5. Secondary Outcome: Minimum Concentration (Cmin) of Emirodatamab
Description: as for outcome 4
Time Frame: as for outcome 4
Population: as for outcome 3
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Cohort 1 (FIH): Emirodatamab Dose A | Cohort 2 (FIH): Emirodatamab Dose B | Cohort 3 (FIH): Emirodatamab Dose C | Cohort 4 (FIH): Emirodatamab Dose D | Cohort 5 (FIH): Emirodatamab Dose E | Cohort 6 (FIH): Emirodatamab Dose F | Cohort 7a (FIH): Emirodatamab Dose G | Cohort 7b (FIH): Emirodatamab Dose F/Dose G | Cohort 8 (FIH): Emirodatamab Dose F/Dose H | Cohort 9 (FIH): Emirodatamab Dose F/Dose H/Dose I | Cohort 10 (FIH): Emirodatamab Dose F/Dose H/Dose J | Cohort 11 (FIH): Emirodatamab Dose F/Dose H/Dose K | Cohort 12 (FIH): Emirodatamab Dose F/Dose H/Dose L | Cohort 13 (FIH): Emirodatamab Dose F/Dose H/Dose M | Cohort 14 (eIV): Emirodatamab Dose F/Dose H/Dose J/Dose K | Cohort 15 (eIV): Emirodatamab Dose F/Dose H/Dose J | Cohort 16: Etanercept + Emirodatamab Dose E | Cohort 17: Etanercept + Emirodatamab Dose F
Number analyzed (Participants) | 1 | 1 | 1 | 0 | 4 | 3 | 1 | 3 | 3 | 4 | 3 | 3 | 5 | 3 | 6 | 1 | 3 | 1
ng/mL
  C1D5 Free Emirodatamab: number analyzed (Participants) | 1 | 1 | 1 | 0 | 4 | 3 | 1 | 3 | 3 | 4 | 3 | 3 | 5 | 3 | 0 | 0 | 3 | 1
  C1D5 Free Emirodatamab | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] |  | 0.00 [0.00 to 0.0569] | 0.00 [0.00 to 0.228] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.149] | 0.0510 [0.00 to 1.42] | 0.434 [0.0833 to 2.79] | 1.10 [0.00 to 3.23] | 0.301 [0.231 to 5.42] | 0.228 [0.00 to 18.5] | 0.00 [0.00 to 16.0] |  |  | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  C1D8 Free Emirodatamab: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 1 | 0 | 0
  C1D8 Free Emirodatamab |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 5.70 [0.00 to 21.6] | 0.253 [0.253 to 0.253] |  |

6. Secondary Outcome: Area Under the Concentration-time Curve (AUC) From Time 0 to Time of Last Quantifiable Concentration (AUC0-last) of Emirodatamab
Description: Serum concentrations of emirodatamab were determined using a validated assay. Noncompartmental analysis was performed for estimation of PK parameters. Concentrations below the LLOQ (0.05 ng/mL) were set to zero before data analysis. AUC(0-last) was calculated using the linear trapezoidal method.
Time Frame: as for outcome 4
Population: as for outcome 3
Measure: Median (Full Range); unit: hour*ng/mL
Arm/Group | Cohort 1 (FIH): Emirodatamab Dose A | Cohort 2 (FIH): Emirodatamab Dose B | Cohort 3 (FIH): Emirodatamab Dose C | Cohort 4 (FIH): Emirodatamab Dose D | Cohort 5 (FIH): Emirodatamab Dose E | Cohort 6 (FIH): Emirodatamab Dose F | Cohort 7a (FIH): Emirodatamab Dose G | Cohort 7b (FIH): Emirodatamab Dose F/Dose G | Cohort 8 (FIH): Emirodatamab Dose F/Dose H | Cohort 9 (FIH): Emirodatamab Dose F/Dose H/Dose I | Cohort 10 (FIH): Emirodatamab Dose F/Dose H/Dose J | Cohort 11 (FIH): Emirodatamab Dose F/Dose H/Dose K | Cohort 12 (FIH): Emirodatamab Dose F/Dose H/Dose L | Cohort 13 (FIH): Emirodatamab Dose F/Dose H/Dose M | Cohort 14 (eIV): Emirodatamab Dose F/Dose H/Dose J/Dose K | Cohort 15 (eIV): Emirodatamab Dose F/Dose H/Dose J | Cohort 16: Etanercept + Emirodatamab Dose E | Cohort 17: Etanercept + Emirodatamab Dose F
Number analyzed (Participants) | 1 | 0 | 1 | 1 | 4 | 3 | 1 | 3 | 3 | 4 | 3 | 3 | 5 | 3 | 6 | 2 | 5 | 1
hour*ng/mL
  C1D5 Free Emirodatamab: number analyzed (Participants) | 1 | 0 | 1 | 1 | 4 | 3 | 1 | 3 | 3 | 4 | 3 | 3 | 5 | 3 | 0 | 0 | 5 | 1
  C1D5 Free Emirodatamab | 0.793 [0.793 to 0.793] |  | 0.484 [0.484 to 0.484] | 0.0894 [0.0894 to 0.0894] | 24.9 [12.1 to 172] | 15.1 [5.89 to 313] | 26.8 [26.8 to 26.8] | 75.5 [38.0 to 1110] | 160 [112 to 1530] | 345 [282 to 3400] | 4590 [122 to 5900] | 611 [384 to 6980] | 1460 [154 to 14100] | 288 [250 to 13100] |  |  | 5.73 [0.962 to 23.7] | 22.6 [22.6 to 22.6]
  C1D8 Free Emirodatamab: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2 | 0 | 0
  C1D8 Free Emirodatamab |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 3550 [60.0 to 11000] | 464 [170 to 758] |  |

7. Secondary Outcome: AUC From Time 0 to Infinity (AUC0-inf) of Emirodatamab
Description: Serum concentrations of emirodatamab were determined using a validated assay. Noncompartmental analysis was performed for estimation of PK parameters. Concentrations below the LLOQ (0.05 ng/mL) were set to zero before data analysis. The AUC(0-inf) was calculated using the linear trapezoidal method.
Time Frame: as for outcome 4
Population: as for outcome 3
Measure: Median (Full Range); unit: hour*ng/mL
Arm/Group | Cohort 1 (FIH): Emirodatamab Dose A | Cohort 2 (FIH): Emirodatamab Dose B | Cohort 3 (FIH): Emirodatamab Dose C | Cohort 4 (FIH): Emirodatamab Dose D | Cohort 5 (FIH): Emirodatamab Dose E | Cohort 6 (FIH): Emirodatamab Dose F | Cohort 7a (FIH): Emirodatamab Dose G | Cohort 7b (FIH): Emirodatamab Dose F/Dose G | Cohort 8 (FIH): Emirodatamab Dose F/Dose H | Cohort 9 (FIH): Emirodatamab Dose F/Dose H/Dose I | Cohort 10 (FIH): Emirodatamab Dose F/Dose H/Dose J | Cohort 11 (FIH): Emirodatamab Dose F/Dose H/Dose K | Cohort 12 (FIH): Emirodatamab Dose F/Dose H/Dose L | Cohort 13 (FIH): Emirodatamab Dose F/Dose H/Dose M | Cohort 14 (eIV): Emirodatamab Dose F/Dose H/Dose J/Dose K | Cohort 15 (eIV): Emirodatamab Dose F/Dose H/Dose J | Cohort 16: Etanercept + Emirodatamab Dose E | Cohort 17: Etanercept + Emirodatamab Dose F
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 3 | 1 | 3 | 3 | 3 | 3 | 3 | 5 | 3 | 6 | 2 | 1 | 1
hour*ng/mL
  C1D5 Free Emirodatamab: number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 3 | 1 | 3 | 3 | 3 | 3 | 3 | 5 | 3 | 0 | 0 | 1 | 1
  C1D5 Free Emirodatamab |  |  |  |  | 26.5 [25.7 to 176] | 16.4 [6.74 to 332] | 28.5 [28.5 to 28.5] | 77.2 [39.3 to 1130] | 169 [114 to 1680] | 314 [290 to 3590] | 4660 [125 to 6220] | 631 [403 to 7410] | 1460 [160 to 15900] | 322 [252 to 14500] |  |  | 17.4 [17.4 to 17.4] | 25.2 [25.2 to 25.2]
  C1D8 Free Emirodatamab: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2 | 0 | 0
  C1D8 Free Emirodatamab |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 3940 [61.4 to 12400] | 473 [178 to 767] |  |

8. Secondary Outcome: AUC From Time Zero to 14 Days Post-dose (AUC14d) of Emirodatamab
Description: Serum concentrations of emirodatamab were determined using a validated assay. Noncompartmental analysis was performed for estimation of PK parameters. Concentrations below the LLOQ (0.05 ng/mL) were set to zero before data analysis. AUC(14d) was calculated as the sum of AUC values of all dosing days in cycle 1.
Time Frame: For all cohorts: from time zero to 14-days following the C1D1 dose (1 cycle= 14 days)
Population: as for outcome 3
Measure: Median (Full Range); unit: hour*ng/mL
Arm/Group | Cohort 1 (FIH): Emirodatamab Dose A | Cohort 2 (FIH): Emirodatamab Dose B | Cohort 3 (FIH): Emirodatamab Dose C | Cohort 4 (FIH): Emirodatamab Dose D | Cohort 5 (FIH): Emirodatamab Dose E | Cohort 6 (FIH): Emirodatamab Dose F | Cohort 7a (FIH): Emirodatamab Dose G | Cohort 7b (FIH): Emirodatamab Dose F/Dose G | Cohort 8 (FIH): Emirodatamab Dose F/Dose H | Cohort 9 (FIH): Emirodatamab Dose F/Dose H/Dose I | Cohort 10 (FIH): Emirodatamab Dose F/Dose H/Dose J | Cohort 11 (FIH): Emirodatamab Dose F/Dose H/Dose K | Cohort 12 (FIH): Emirodatamab Dose F/Dose H/Dose L | Cohort 13 (FIH): Emirodatamab Dose F/Dose H/Dose M | Cohort 14 (eIV): Emirodatamab Dose F/Dose H/Dose J/Dose K | Cohort 15 (eIV): Emirodatamab Dose F/Dose H/Dose J | Cohort 16: Etanercept + Emirodatamab Dose E | Cohort 17: Etanercept + Emirodatamab Dose F
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 4 | 3 | 1 | 3 | 3 | 4 | 3 | 3 | 5 | 3 | 6 | 2 | 5 | 1
hour*ng/mL | 0.454 [0.454 to 0.454] | 0.0401 [0.0401 to 0.0401] | 0.323 [0.323 to 0.323] | 0.377 [0.377 to 0.377] | 52.8 [2.93 to 262] | 28.8 [13.3 to 523] | 48.0 [48.0 to 48.0] | 103 [59.2 to 1470] | 237 [139 to 1770] | 518 [103 to 4890] | 5320 [155 to 7210] | 762 [489 to 9250] | 1670 [215 to 17700] | 374 [293 to 15300] | 5070 [163 to 17400] | 923 [676 to 1170] | 4.52 [0.434 to 38.2] | 44.3 [44.3 to 44.3]

9. Secondary Outcome: Terminal Half-life (t1/2,z) of Emirodatamab
Description: Serum concentrations of emirodatamab were determined using a validated assay. Noncompartmental analysis was performed for estimation of PK parameters. Concentrations below the LLOQ (0.05 ng/mL) were set to zero before data analysis. t1/2,z was calculated as t1/2,z = ln(2)/λz, where λz is the first-order terminal rate constant estimated via linear regression of the terminal log-linear phase.
Time Frame: as for outcome 4
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1 (FIH): Emirodatamab Dose A | Cohort 2 (FIH): Emirodatamab Dose B | Cohort 3 (FIH): Emirodatamab Dose C | Cohort 4 (FIH): Emirodatamab Dose D | Cohort 5 (FIH): Emirodatamab Dose E | Cohort 6 (FIH): Emirodatamab Dose F | Cohort 7a (FIH): Emirodatamab Dose G | Cohort 7b (FIH): Emirodatamab Dose F/Dose G | Cohort 8 (FIH): Emirodatamab Dose F/Dose H | Cohort 9 (FIH): Emirodatamab Dose F/Dose H/Dose I | Cohort 10 (FIH): Emirodatamab Dose F/Dose H/Dose J | Cohort 11 (FIH): Emirodatamab Dose F/Dose H/Dose K | Cohort 12 (FIH): Emirodatamab Dose F/Dose H/Dose L | Cohort 13 (FIH): Emirodatamab Dose F/Dose H/Dose M | Cohort 14 (eIV): Emirodatamab Dose F/Dose H/Dose J/Dose K | Cohort 15 (eIV): Emirodatamab Dose F/Dose H/Dose J | Cohort 16: Etanercept + Emirodatamab Dose E | Cohort 17: Etanercept + Emirodatamab Dose F
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 3 | 1 | 3 | 3 | 3 | 3 | 3 | 5 | 3 | 6 | 2 | 1 | 1
hours
  C1D5 Free Emirodatamab: number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 3 | 1 | 3 | 3 | 3 | 3 | 3 | 5 | 3 | 0 | 0 | 1 | 1
  C1D5 Free Emirodatamab |  |  |  |  | 23.9 [10.2 to 49.7] | 25.5 [8.29 to 55.3] | 14.1 [14.1 to 14.1] | 28.1 [14.9 to 52.9] | 45.0 [19.3 to 75.7] | 39.0 [26.2 to 46.9] | 42.1 [13.9 to 68.5] | 53.0 [46.3 to 56.9] | 40.4 [12.4 to 66.2] | 32.3 [11.1 to 57.4] |  |  | 12.4 [12.4 to 12.4] | 20.8 [20.8 to 20.8]
  C1D8 Free Emirodatamab: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2 | 0 | 0
  C1D8 Free Emirodatamab |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 38.0 [9.05 to 62.6] | 22.7 [19.8 to 25.5] |  |

10. Secondary Outcome: Best Overall Response According to Revised International Working Group (IWG) Response Criteria
Description: A response consisted of any of the following, assessed according to the IWG response criteria:
  * complete remission (CR): bone marrow (BM) blasts <5%; no blasts with Auer rods; no extramedullary disease; absolute neutrophil count >1.0 x 10^9/L; platelet count > 100 x 10^9/L; independence of red cell transfusions
  * CR with incomplete recovery of peripheral blood counts (CRi): CR except for residual neutropenia (< 1.0 x 10^9/L) or thrombocytopenia (< 100 x 10^9/L)
  * complete response/remission with partial hematologic recovery (CRh): ≤5% BM blasts, no circulating blasts/extramedullary disease and partial recovery of peripheral blood counts (platelets > 50,000/µL, hemoglobin ≥7g/dL and absolute neutrophil count > 500/µL).
  * morphologic leukemia-free state: BM blasts < 5%; no blasts with Auer rods; no extramedullary disease; no hematologic recovery required
  * partial remission: hematological criteria of CR; decrease BM blast to 5-25%; decrease of pretreatment BM blast percentage by ≤ 50%
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (FIH): Emirodatamab Dose A | Cohort 2 (FIH): Emirodatamab Dose B | Cohort 3 (FIH): Emirodatamab Dose C | Cohort 4 (FIH): Emirodatamab Dose D | Cohort 5 (FIH): Emirodatamab Dose E | Cohort 6 (FIH): Emirodatamab Dose F | Cohort 7a (FIH): Emirodatamab Dose G | Cohort 7b (FIH): Emirodatamab Dose F/Dose G | Cohort 8 (FIH): Emirodatamab Dose F/Dose H | Cohort 9 (FIH): Emirodatamab Dose F/Dose H/Dose I | Cohort 10 (FIH): Emirodatamab Dose F/Dose H/Dose J | Cohort 11 (FIH): Emirodatamab Dose F/Dose H/Dose K | Cohort 12 (FIH): Emirodatamab Dose F/Dose H/Dose L | Cohort 13 (FIH): Emirodatamab Dose F/Dose H/Dose M | Cohort 14 (eIV): Emirodatamab Dose F/Dose H/Dose J/Dose K | Cohort 15 (eIV): Emirodatamab Dose F/Dose H/Dose J | Cohort 16: Etanercept + Emirodatamab Dose E | Cohort 17: Etanercept + Emirodatamab Dose F
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 5 | 4 | 2 | 3 | 4 | 4 | 4 | 4 | 7 | 3 | 7 | 3 | 6 | 4
Participants
  CR | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  CRi | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  CRh | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Morphologic leukemia-free state | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 4 | 1 | 0 | 0
  Partial remission | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Treatment failure | 1 | 1 | 1 | 1 | 5 | 4 | 1 | 3 | 3 | 3 | 3 | 2 | 3 | 1 | 2 | 2 | 6 | 2
  No evaluable response | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 2

ADVERSE EVENTS:
Time Frame: For all-cause mortality, from enrollment to end of study; median time on study was 1.347 months. Adverse events were reported from first dose of investigational product (day 1 cycle 1) to 30 days after last dose of investigational product or end of study; median treatment duration was 0.62 months.
Description: All-cause mortality is reported for all participants enrolled in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of trial drug.
Groups:
- Overall Studies: All participants included in all cohorts.
Arm/Group | Cohort 1 (FIH): Emirodatamab Dose A | Cohort 2 (FIH): Emirodatamab Dose B | Cohort 3 (FIH): Emirodatamab Dose C | Cohort 4 (FIH): Emirodatamab Dose D | Cohort 5 (FIH): Emirodatamab Dose E | Cohort 6 (FIH): Emirodatamab Dose F | Cohort 7a (FIH): Emirodatamab Dose G | Cohort 7b (FIH): Emirodatamab Dose F/Dose G | Cohort 8 (FIH): Emirodatamab Dose F/Dose H | Cohort 9 (FIH): Emirodatamab Dose F/Dose H/Dose I | Cohort 10 (FIH): Emirodatamab Dose F/Dose H/Dose J | Cohort 11 (FIH): Emirodatamab Dose F/Dose H/Dose K | Cohort 12 (FIH): Emirodatamab Dose F/Dose H/Dose L | Cohort 13 (FIH): Emirodatamab Dose F/Dose H/Dose M | Cohort 14 (eIV): Emirodatamab Dose F/Dose H/Dose J/Dose K | Cohort 15 (eIV): Emirodatamab Dose F/Dose H/Dose J | Cohort 16: Etanercept + Emirodatamab Dose E | Cohort 17: Etanercept + Emirodatamab Dose F | Overall Studies
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/1 | 1/5 | 1/4 | 0/2 | 2/3 | 1/4 | 2/4 | 1/4 | 0/4 | 2/7 | 1/3 | 1/7 | 1/3 | 0/6 | 1/4 | 14/64
Serious Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 0/1 | 0/1 | 3/5 | 4/4 | 2/2 | 1/3 | 1/4 | 2/4 | 4/4 | 2/4 | 5/7 | 2/3 | 5/7 | 2/3 | 2/6 | 3/4 | 40/64
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/1 | 1/1 | 5/5 | 4/4 | 2/2 | 3/3 | 4/4 | 4/4 | 4/4 | 4/4 | 7/7 | 3/3 | 7/7 | 3/3 | 6/6 | 4/4 | 64/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (FIH): Emirodatamab Dose A (N=1) | Cohort 2 (FIH): Emirodatamab Dose B (N=1) | Cohort 3 (FIH): Emirodatamab Dose C (N=1) | Cohort 4 (FIH): Emirodatamab Dose D (N=1) | Cohort 5 (FIH): Emirodatamab Dose E (N=5) | Cohort 6 (FIH): Emirodatamab Dose F (N=4) | Cohort 7a (FIH): Emirodatamab Dose G (N=2) | Cohort 7b (FIH): Emirodatamab Dose F/Dose G (N=3) | Cohort 8 (FIH): Emirodatamab Dose F/Dose H (N=4) | Cohort 9 (FIH): Emirodatamab Dose F/Dose H/Dose I (N=4) | Cohort 10 (FIH): Emirodatamab Dose F/Dose H/Dose J (N=4) | Cohort 11 (FIH): Emirodatamab Dose F/Dose H/Dose K (N=4) | Cohort 12 (FIH): Emirodatamab Dose F/Dose H/Dose L (N=7) | Cohort 13 (FIH): Emirodatamab Dose F/Dose H/Dose M (N=3) | Cohort 14 (eIV): Emirodatamab Dose F/Dose H/Dose J/Dose K (N=7) | Cohort 15 (eIV): Emirodatamab Dose F/Dose H/Dose J (N=3) | Cohort 16: Etanercept + Emirodatamab Dose E (N=6) | Cohort 17: Etanercept + Emirodatamab Dose F (N=4) | Overall Studies (N=64)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 7
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 1 | 0 | 0 | 10
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bacillus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Enterobacter bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fungal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mucormycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neutropenic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 4
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Post procedural cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Puncture site cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 4
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Sinusitis fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 5
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (FIH): Emirodatamab Dose A (N=1) | Cohort 2 (FIH): Emirodatamab Dose B (N=1) | Cohort 3 (FIH): Emirodatamab Dose C (N=1) | Cohort 4 (FIH): Emirodatamab Dose D (N=1) | Cohort 5 (FIH): Emirodatamab Dose E (N=5) | Cohort 6 (FIH): Emirodatamab Dose F (N=4) | Cohort 7a (FIH): Emirodatamab Dose G (N=2) | Cohort 7b (FIH): Emirodatamab Dose F/Dose G (N=3) | Cohort 8 (FIH): Emirodatamab Dose F/Dose H (N=4) | Cohort 9 (FIH): Emirodatamab Dose F/Dose H/Dose I (N=4) | Cohort 10 (FIH): Emirodatamab Dose F/Dose H/Dose J (N=4) | Cohort 11 (FIH): Emirodatamab Dose F/Dose H/Dose K (N=4) | Cohort 12 (FIH): Emirodatamab Dose F/Dose H/Dose L (N=7) | Cohort 13 (FIH): Emirodatamab Dose F/Dose H/Dose M (N=3) | Cohort 14 (eIV): Emirodatamab Dose F/Dose H/Dose J/Dose K (N=7) | Cohort 15 (eIV): Emirodatamab Dose F/Dose H/Dose J (N=3) | Cohort 16: Etanercept + Emirodatamab Dose E (N=6) | Cohort 17: Etanercept + Emirodatamab Dose F (N=4) | Overall Studies (N=64)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 2 | 2 | 10
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 8
Hypofibrinogenaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 4
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 4
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Aortic valve disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Mitral valve disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 5
Tricuspid valve disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Asthenopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Exophthalmos (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Eye irritation (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 8
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 3 | 1 | 1 | 3 | 0 | 0 | 0 | 13
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 4 | 1 | 2 | 0 | 15
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 5
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Lip pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Mouth swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 2 | 2 | 1 | 1 | 2 | 3 | 0 | 0 | 0 | 15
Oral mucosal erythema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 3
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 5
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Rectal discharge (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Reflux gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 3
Tooth erosion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 8
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 9
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 2 | 0 | 1 | 1 | 0 | 2 | 1 | 1 | 0 | 13
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 1 | 1 | 0 | 12
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 7
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Physical deconditioning (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 3
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 3 | 2 | 2 | 0 | 1 | 1 | 1 | 15
Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Swelling face (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 3
Temperature intolerance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Periportal oedema (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 4 | 2 | 2 | 3 | 4 | 4 | 4 | 4 | 6 | 3 | 7 | 2 | 5 | 2 | 52
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alpha haemolytic streptococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 4
Bacteroides bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colonic abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cystitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device related bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Enterobacter bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Enterococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Escherichia infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Perirectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Respiratory tract infection fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Sinusitis fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Peripancreatic fluid collection (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 1 | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 12
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Antithrombin III decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 3 | 0 | 10
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Blood fibrinogen decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 3
Blood urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Lipase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 6
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 0 | 6
Transaminases (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Appetite disorder (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 4
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 3
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 7
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 8
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 3 | 3 | 1 | 0 | 4 | 2 | 1 | 0 | 19
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 3 | 1 | 2 | 2 | 1 | 1 | 0 | 16
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 0 | 2 | 0 | 0 | 0 | 11
Hypouricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 0 | 0 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3 | 1 | 3 | 1 | 0 | 0 | 0 | 11
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Central nervous system lesion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 4
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Formication (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 1 | 1 | 3 | 0 | 1 | 1 | 0 | 0 | 12
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 4
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Myoclonus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 3
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 5
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Nightmare (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Restlessness (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urethral pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Penile pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 9
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 6
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 6
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 4
Pulmonary hilum mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Nail bed bleeding (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 8
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 8
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 6
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Due to the early termination of the study, the dose expansion cohort was not opened, and the secondary endpoint for duration of response which was pre-specified for the dose expansion cohort was not collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2022-03-16): https://cdn.clinicaltrials.gov/large-docs/69/NCT03541369/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/69/NCT03541369/SAP_001.pdf